CLINICAL TRIAL: NCT07000877
Title: Nasal Decongestant Administration to Reduce Perioperative Adverse Events in Children With Upper Respiratory Track Infections Having General Anesthesia - a Low Risk Intervention. (NARWHAL)
Brief Title: Nasal Decongestant to Reduce Perioperative Adverse Events in Children With Upper Respiratory Track Infections Having Anesthesia.
Acronym: NARWHAL
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Telethon Kids Institute (Other)
Collaborators: Child and Adolescent Health Service - Perth (Other Government); Hospital das Clínicas de São Paulo - SP (Unknown); Rigshospitalet, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: RGS0000007387
Record Dates: First submitted 2025-05-13; First posted 2025-06-03 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-09

CONDITIONS: Perioperative Respiratory Adverse Events; Anesthesia Outcomes
Keywords: perioperative respiratory adverse events; nasal decongestant; upper respiratory tract infection; Children; surgery; pediatrics; anesthesia
MeSH Terms: conditions — Respiratory Tract Infections | interventions — Oxymetazoline; Saline Solution

STUDY DESIGN:
Intervention Model Description: Multicentre, double-blinded randomised controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double Blind trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Decongestant nasal spray (oxymetazoline hydrochloride 0.05%) (Active Comparator): Decongestant nasal spray, oxymetazoline (0.05%). Specific: 2.5mL of oxymetazoline 0.05% dispensed into amber brown 15ml bottles with pump and actuator attached. Children aged 1 to 5.99 years will receive 1 spray of either the nasal decongestant or placebo into each nostril, while children aged 6 years and above will receive 2 spays per nostril. Administration will be recorded on the standard patient's Medication Chart.
  Interventions: Drug: Decongestant nasal spray (oxymetazoline hydrochloride (0.05%))
- Placebo Comparator : Placebo spray (control group) (Placebo Comparator): Matched Placebo spray. Specific: 2.5mL of normal saline 0.9% and benzalkonium chloride 0.02% dispensed into amber brown 15ml bottles with pump and actuator attached. Dose: children aged 1 to 5.99 years will receive 1 spray of either the nasal decongestant or placebo into each nostril, while children aged 6 years and above will receive 2 spays per nostril. Administration will be recorded on the standard patient's Medication Chart.
  Interventions: Drug: PLACEBO: 2.5mL of normal saline 0.9% and benzalkonium chloride 0.02%

INTERVENTIONS:
Drug: Decongestant nasal spray (oxymetazoline hydrochloride (0.05%)) — Decongestant nasal spray containing active ingredient.
  Arms: Decongestant nasal spray (oxymetazoline hydrochloride 0.05%)
Drug: PLACEBO: 2.5mL of normal saline 0.9% and benzalkonium chloride 0.02% — Control nasal spray containing no active ingredient.
  Arms: Placebo Comparator : Placebo spray (control group)

SUMMARY:
The goal of this multicentre, double-blind, randomised controlled trial study is to learn if the use of a nasal spray to open the nasal passages and increase airflow before surgery can reduce the occurrence of perioperative respiratory adverse events in children with upper respiratory tract infection who are undergoing anesthesia.

The main questions it aims to answer are:

* Does use of a nasal decongestant (Oxymetazoline 0.05%) reduce perioperative respiratory adverse events during emergence (when waking up from anesthesia) or in the post-anesthesia care unit in children.
* Is it easy and acceptable to doctors, children and parents to use the nasal decongestant treatment? Researchers will compare the nasal decongestant to a placebo (a look-alike substance that contains no drug) to see if it works to reduce perioperative respiratory adverse effects.

Participants will:

* Take a nasal decongestant or a placebo prior to surgery (just before anaesthesia is given)
* Be monitored during and after surgery in the post-anaesthesia care unit for any perioperative respiratory adverse events.
* Be asked about how acceptable they found the treatment.

DETAILED DESCRIPTION:
Upper respiratory tract infections (URTI), including COVID-19 infection and the common cold, are common and frequent in children who present for elective surgery. Children with URTI are at a two-to-three-fold increased risk of perioperative respiratory adverse events (PRAE). PRAE are among the most serious and impactful consequences of paediatric anesthesia, including cardio-respiratory arrest, and therefore present a significant challenge for the pediatric anesthetist.

This two-phase, multicentre, international, double-blinded, randomised controlled trial aims to improve the safety of children with upper respiratory tract infections undergoing anesthesia by investigating the use of a nasal spray pre-operatively to reduce respiratory complications. Following informed written parental consent, 200 pediatric patients aged 1 to 8 years, undergoing general anesthesia for any surgery with current or recent URTI will be randomised to receive at the induction of anesthesia either a decongestant nasal spray or a placebo spray using the same bottle/actuator.

Monitoring and recording of PRAE (laryngospasm - closure of the vocal cords, bronchospasm - narrowing of the airways, severe and persistent coughing, airway obstruction, oxygen desaturation (<95%) and postoperative stridor-squeaky noises when breathing) will occur throughout the procedure and in the post anesthesia care unit (PACU). We hypothesise that children who receive the nasal decongestant will be at a reduced risk of developing PRAE.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 1 to 8.99 years with a current or recent upper respiratory tract infection (<2 weeks).
* Undergoing interventions or surgery under general anesthesia (elective or urgent not emergency).

Exclusion Criteria:

* Currently taking nasal decongestants (past 24 hours) or receiving co-phenylocaine or decongestion for surgery.
* Surgery impacting the nasal airflow, e.g. adenoidectomy, cautery of inferior turbinates.
* Airway management with an endotracheal tube, face mask or high flow nasal oxygen.
* Known cardiovascular, respiratory or neurological disorders giving an ASA III or above.
* Thyroid disease.
* Diabetes.
* Known hypersensitivity to the interventional products.
* Department of Child Protection and Family Services involved in their care.
* Planned admissions to the Paediatric Intensive Care Unit (PICU).

Ages: 1 Year to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2025-06-25 (Actual); Primary Completion 2028-05-30 (Estimated); Study Completion 2028-05-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of perioperative respiratory adverse event (PRAE) following the delivery of a nasal decongestant (Oxymetazoline 0.05%) or placebo prior to surgery under anesthesia in children with upper respiratory tract infection | On day of surgery: Perioperative period. PRAE will be assessed if it occurs anywhere along the perioperative pathway between the beginning of the patient's emergence from anesthesia and their discharge from the post-anesthetic care unit (PACU)
  PRAE will be defined as laryngospasm, bronchospasm, severe persistant coughing, hypoxaemia (<95% for at least 10 seconds), airway obstruction, stridor or pulmonary aspiration. Incidence will be assessed by the clinician caring for the patient. Incidence is binary - yes if PRAE occured, no otherwise.

SECONDARY OUTCOMES:
Assess the incidence of severe PRAE during emergence or in PACU in children who received the decongestant spray compared to the control group. | Day of surgery: Perioperative period. Severe PRAE will be assessed if it occurs anywhere along the perioperative pathway between the beginning of the patient's emergence from anesthesia and their discharge from the post-anesthetic care unit (PACU)
  Severe PRAE is defined as laryngospasm or bronchospasm, as assessed by the clinician caring for the patient.
Assess the incidence of minor PRAE during emergence or in PACU inchildren who recieved the decongestant spray compared to the control group. | Day of surgery: Perioperative period. Minor PRAE will be assessed if it occurs anywhere along the perioperative pathway between the beginning of the patient's emergence from anesthesia and their discharge from the post-anesthetic care unit (PACU)
  Minor PRAE is defined as severe coughing, desaturation <95% for at least 10 seconds, airway obstruction, stridor or pulmonary aspiration, as assessed by the clinician caring for the patient.
Evaluate the acceptability of nasal decongestant use at the induction of anesthesia in children with upper respiratory tract infection aged 4 and older and their parents/guardians | Patients and parents/guardians will be asked to rate the intervention post-operatively, prior to their discharge from hospital.
  Children aged 4 and over and their parents/guardians will be asked to rate the acceptibility of the intervention using a 5-point Likert scale (1 = completely unacceptable; 5 = completely acceptable).
Evaluate the acceptability of nasal decongestant use at the induction of anesthesia by the treating anaesthetist | Treating anaesthetists will be asked to rate the intervention immediately after the administration of the interventional product.
  Treating anaesthetists will be asked to rate the acceptibility of the intervention on a 5-point Likert scale (1 = completely unacceptable; 5 = completely acceptable)
Incidence of any potential adverse effects related to the administration of the nasal decongestant/placebo | Any potential adverse effects will be assessed from the administration of the interventional product until the patient's discharge from hospital.
  Any potential adverse effects will be recorded as per the study doctor and the clinical team caring for the patient.
Assessment of the successful administration of the interventional product in children | Successful administration of the interventional product will be assessed by the study team at induction of anesthesia, immediately following the administration or attempted administration of the nasal decongestant or placebo.
  This will be based upon the clinical judgement of the treating anesthesia clinician.

CONTACTS AND LOCATIONS:
Locations (1):
- Perth Children's Hospital, Perth, We, Australia

IPD SHARING:
Plan to Share IPD: No